CLINICAL TRIAL: NCT05182437
Title: Precision Radiation Treatment for Epilepsy (PRECISION)
Acronym: PRECISION
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other); UMC Utrecht (Other); Amsterdam University Medical Center (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80-86200-98- 25008
Record Dates: First submitted 2021-09-27; First posted 2022-01-10 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial Observational Model : Experimental Time Perspective : Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LINAC-based Stereotactic Radiotherapy (Experimental): The intervention will consist of a single LINAC based SRT treatment and is given by the radiation-oncologist after detailed localisation of the epileptogenic zone (EZ) with the neurologist, radiologist and neurosurgeon.
  Interventions: Radiation: LINAC-based Stereotactic Radiotherapy
- Randomised waitlist-controlled trial (Other): The first 2 years after randomization stardard treatment (AED continuation and neuromodulation). After 2-year follow up the waitlist-control group, patients are offered the intervention (LINAC-based Stereotactic Radiotherapy). This intervention is optional
  Interventions: Radiation: LINAC-based Stereotactic Radiotherapy

INTERVENTIONS:
Radiation: LINAC-based Stereotactic Radiotherapy — Target definition: the target volume is defined as the epileptogenic zone (EZ) on all (non) invasive examinations (e.g. 3, 7 Tesla MRI or Stereo-EEG) of the presurgical path. Planning target volume (PTV) = GTV. A single fraction SRT with a prescribed isotoxic dose of 24 Gy to the 100% surrounding isodose. Dose is depending on the proximity and maximum tolerable dose to the radiosensitive organs at risk and EZ volume resulting in a V12<= 10 cc reducing the risk on radionecrosis.

SUMMARY:
The PRECISION-study offers a non-invasive, curative intervention for drug-resistant localised epilepsy patients who are not eligible for surgery. The intervention will consist of a single LINAC based SRT treatment and is given by the radiation-oncologist after detailed localisation of the epileptogenic zone with the neurologist, radiologist and neurosurgeon.

This intervention will make curative-intent treatment possible where this could otherwise not be given and is a non-invasive and non-competitive alternative to epilepsy surgery. It is expected that the health costs for this curative treatment will not exceed standard treatment, such as lifelong medication and neuromodulation.

DETAILED DESCRIPTION:
In this PRECISION-study including adult patients with drug-resistant, localised epilepsy, not eligible for surgery, we offer non-invasive linear accelerator (LINAC) based Stereotactic Radiotherapy (SRT) with curative intent.

SRT and stereotactic radio-surgery (SRS) have been used to treat several types of neoplasms in the brain for several decades. Several publications (level 2 evidence) have shown the potential value of SRT in patients with drug-resistant epilepsy, however no level-1 evidence was given enabling guideline development. A recent systematic review from our institution has shown that SRT resulted in a significant seizure cure or reduction in 58% of the 170 included patients, within 2 years after treatment. Interestingly, the ROSE trial, randomising between open surgery and SRT, has demonstrated a seizure remission of 52% in the radiotherapy group after 2 years with the proportion of seizure-free patients still increasing with a longer follow-up up to 74% after 3 years. Therefore, SRT may be considered a curative treatment for drug resistant localised epilepsy. Currently, randomized controlled SRT epilepsy trials are lacking and there is a need for high quality evidence, so SRT can be clinically implemented for localised drug-resistant epilepsy patients in the Netherlands as well.

The PRECISION-study is a randomised waitlist-controlled trial in which SRT is the intervention and AED continuation and neuromodulation are the standard treatment with a 1:1 randomization. After 2-year follow up the waitlist-control group, patients are offered the intervention (optional).

We hypothesize that SRT alters the epileptogenic cerebral tissue to yield a reduction in seizures and possibly cure after 2 years, with a significant increase in the patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations
3. Willingness to use contraception by a method that is deemed effective by the Investigator during the SRT treatment and for at least 30 days following the SRT therapy
4. The patient or caretaker is able to keep an epilepsy diary
5. The patient has a diagnosis of epilepsy established by a dedicated neurologist
6. The patient had at least 3 focal-onset seizures over a 3-month period despite two or more antiepileptic medication trials (according ILAE Task Force on therapeutic strategies)
7. Video electroencephalography and work-up in the epilepsy surgery working group to determine a well-circumscribed seizure focus is available
8. Evidence (e.g. 3T-MRI or a clear SEEG delineation) of the anatomic region to be targeted with SRT, correlating with the EZ hypothesis;
9. A functional MRI to lateralize language or localize visual, motor and/or sensory eloquent cortex has been performed in selected patients (if the lesion is expected to be located, based on anatomy, in the language areas).
10. The patient has completed a standard battery of neuropsychological testing
11. The patient been deemed an appropriate candidate for stereotactic radiosurgery by a dedicated Radiation Oncologist and Neurosurgeon/Epileptologist and referred for the study by one of the Dutch regional multidisciplinary epilepsy surgery working groups
12. Patients that were rejected for surgery in an earlier stage can participate in the trial if the last change of the NVS/DBS settings were more than 1 year ago or NVS/DBS was not (yet) tried.

Exclusion Criteria:

1. Pregnancy
2. If a radiation treatment plan without exceeding the constraints for the organs at risk is not feasible.
3. Prior cranial radiotherapy
4. If radiotherapy treatment is not possible for diverse reasons.
5. If the subject has clinically significant and uncontrolled major other medical condition(s) including but not limited to:

ii. psychiatric illness/social situation that would limit compliance with study requirements iii. any medical condition, with the opinion of the study investigator, places the subject at an unacceptably high risk for toxicities iv. Progressive co-morbidity which limits overall survival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Radiotherapy adapted Engel classification (RAEC) is I, II or III | Baseline (before treatment), 1 year, 2 year, 3 year, 4 year and 5 year after treatment
  Radiotherapy adapted Engel classification (RAEC). For analysis of outcomes in the incidence of seizures, we use in this study the Engel classification, adapted for radiotherapy. This includes four classes: class I - seizure free, class II - rarely seizures, class III improved, more than 75% IV- no significant improvement.

SECONDARY OUTCOMES:
Seizure frequency | Baseline (before treatment), 1 year, 2 year, 3 year, 4 year and 5 year after treatment
  self-reports and reports from caretakers, combined in a digital diary.
Seizure-free days | Baseline (before treatment), 1 year, 2 year, 3 year, 4 year and 5 year after treatment
  self-reports and reports from caretakers, combined in a digital diary.
Type of epilepsy | Baseline (before treatment), 1 year, 2 year, 3 year, 4 year and 5 year after treatment
  self-reports and reports from caretakers, combined in a digital diary.
EQ-5D 5 Level (EQ-5D-5L) | Baseline (before treatment), 1 year, 2 year, 3 year, 4 year and 5 year after treatment
  EQ-5D-5L is comprised of a descriptive system and a visual analogue scale. The descriptive system measures quality of life along five dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with five levels for each dimension from which subjects are asked to select one. There are 5 questions and 5 qualitative answers plus a numerical scale (from 0 to 100) related with the general health status. We will attribute a numerical value to the 5 qualitative answers (100 for the best/ 75, 50, 25 and 0 for the worse).
The Assessment of Quality of Life-8 Dimensions Score (AQoL-8D Score) | Baseline (before treatment), 1 year, 2 year, 3 year, 4 year and 5 year after treatment
  The Assessment of Quality of Life (AQoL) measure of health-related Quality of Life. AQoL-8D covers dimensions of Independent Living, Happiness, Mental Health Coping, Relationships, Self-Worth, Pain, and Senses. Items are scored from 0 to 3. Scores range from 0 to 45 with higher scores indicating poorer quality of life
Quality of life in Epilepsy-31 Inventory (QOLIE-31) | Baseline (before treatment), 1 year, 2 year, 3 year, 4 year and 5 year after treatment
  The QOLIE includes 31 questions about health and daily activities. Responses are given on a range of scales. Responses are coded to 0 to 100 point scales where higher scores indicate better quality of life. The final score is the average of scores for the individual items.
  QOLIE-31 is a widely used epilepsy-specific questionnaire
'Cost-effectiveness Resource use' is measured with iMTA Productivity Cost Questionnaire (iPCQ) | Baseline (before treatment), 1 year, 2 year, 3 year, 4 year and 5 year after treatment
  Institute for Medical Technology Assessment (iMTA) Productivity Cost Questionnaire (iPCQ). The iPCQ is a standardized instrument for measuring and valuing health related productivity losses. This wil be used for the cost effectiveness analysis.
'Cost-effectiveness Resource use' is measured with iMTA Medical Consumption Questionnaire (iMCQ) | Baseline (before treatment), 1 year, 2 year, 3 year, 4 year and 5 year after treatment
  Institute for Medical Technology Assessment (iMTA) Medical Consumption Questionnaire (iMCQ). The iMCQ is a standardized instrument for measuring medical costs.
  The aim of the iVICQ is to facilitate and promote an accurate description of providing informal care, its effects on informal caregivers, and how such effects are included in economic evaluations of health care interventions.
'Informal care' is meausured with iMTA Valuation of Informal Care Questionnaire (iVICQ) | Baseline (before treatment), 1 year, 2 year, 3 year, 4 year and 5 year after treatment
  Institute for Medical Technology Assessment (iMTA) Valuation of Informal Care Questionnaire (iVICQ).
  The aim of this standardized instrument is to facilitate and promote an accurate description of providing informal care, its effects on informal caregivers, and how such effects are included in economic evaluations of health care interventions.
'Patients' experiences' are measured with the instrument 'Patient Reported Experience Measures Medical Specialtic Care' (PREM MSZ) Medical Specialistic Care (PREM MSZ) | Baseline (before treatment), 1 year, 2 year, 3 year, 4 year and 5 year after treatment
  PREM MSZ is a Dutch standardized questionnaire to report Patient Reported Experience. Instrument is developed by NIVEL (Dutch Institute for Healthcare Research) in collabaration with Dutch healcare insurers. Instrument includes 13 questions about the satisfaction with the communication between the patient and the caregiver, shared decision making, trust in the expertise of the physician, the effect of the treatment. Responses to these questions are coded into 0 to 10 points. Higher scores indicate higher satisfaction with care. In the questionnaire patients are also asked for the evaluation of their own health, recommendations to improve care, and if they would recommend the care to other patients with the same health problem. Finally there are some questions about background variables (age, gender, education)

CONTACTS AND LOCATIONS:
Overall Officials: Daniëlle Eekers, Dr., Principal Investigator — Radiation Oncologist
Locations (1):
- Maastricht Radiation Oncology, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eekers DBP, Pijnappel EN, Schijns OEMG, Colon A, Hoeben A, Zindler JD, Postma AA, Hoffmann AL, Lambin P, Troost EGC. Evidence on the efficacy of primary radiosurgery or stereotactic radiotherapy for drug-resistant non-neoplastic focal epilepsy in adults: A systematic review. Seizure. 2018 Feb;55:83-92. doi: 10.1016/j.seizure.2018.01.009. Epub 2018 Jan 31. PMID 29414140
- [Derived] Zegers CML, Swinnen A, Roumen C, Hoffmann AL, Troost EGC, van Asch CJJ, Brandts L, Compter I, Dieleman EMT, Dijkstra JB, Granzier M, Hendriks M, Hofman P, Houben RMA, Ramaekers B, Ronner HE, Rouhl RPW, van der Salm S, Santegoeds RGC, Verhoeff JJ, Wagner GL, Zwemmer J, Schijns O, Colon AJ, Eekers DBP. High-precision stereotactic irradiation for focal drug-resistant epilepsy versus standard treatment: a randomized waitlist-controlled trial (the PRECISION trial). Trials. 2024 May 21;25(1):334. doi: 10.1186/s13063-024-08168-9. PMID 38773643
- See also: Publication Pubmed — https://pubmed.ncbi.nlm.nih.gov/29414140/